CLINICAL TRIAL: NCT05429255
Title: Aerobic Training vs Exergame Training in Patients With Chronic Mild-Moderate Stroke
Brief Title: Aerobic Exercise in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU0558
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Aerobic; Exergame
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: Person performing outcome assessments will not know which group the patient is assigned. Participant cannot be blinded given nature of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training (Experimental): Participants will be given a stationary exercise bike for home use. They will be instructed to use the exercise bike five times a week for thirty-minute sessions. The exercise intensity prescription will be based on the subject's maximum heart rate based on age. The exercise program will start at 60% of max heart rate, and then will be increased by steps of 5% intensity every 2 weeks until participants reach 30 minutes of training at 80% intensity. In addition, rate of perceived exertion (Borg scale) will be assessed at each training session. Participants will be contacted weekly by email or phone to answer any questions about the exercise protocol and will be instructed to log each training session.
  Subjects will record duration of exercise, perceived exertion, average heart rate, maximum heart rate, and distance.
  Subjects will be asked to use the bike for 1 month
  Interventions: Behavioral: Aerobic Exercise
- Exergame Training (Active Comparator): The Nintendo wii system will be used as the rehabilitation exergame system in the study. Wii-fit games will be used and the subjects will be shown to system at the initial assessment. Participants will be instructed to play 30 minutes a day, 5 days per week for 1 month. Participants will be contacted weekly by email or phone to answer any questions about the exercise protocol and will be instructed to log each training session.
  Subjects will record duration of exercise, perceived exertion, balance challenge, and which games they played.
  Interventions: Behavioral: Exergame Training

INTERVENTIONS:
Behavioral: Aerobic Exercise — Bicycle training
  Arms: Aerobic Training
Behavioral: Exergame Training — Nintendo Wii
  Arms: Exergame Training

SUMMARY:
The purpose of this study is to compare aerobic training to exergame training in people with chronic mild/moderate stroke. The objectives of this study are two-fold: 1) To evaluate the effects of a home-based aerobic exercise cycle ergometer program on cardiorespiratory fitness, mobility, cognitive, and exercise self-efficacy outcomes in subacute and chronic stroke patients; and 2) to evaluate the effects of an exergaming program on the same outcomes.

DETAILED DESCRIPTION:
Annually, 13.7 million strokes occur worldwide, placing it as a leading cause of death and disability, especially among older adults. Stroke survivors often face significant cognitive and motor impairments for months to years after a stroke event, creating significant deficits in functional capacity during activities of daily living (ADLs), as well as in overall quality of life. Stroke patients have identified interventions to improve cognitive outcomes, mobility training, and exercise programs as top priorities for guiding research pursuits.

Aerobic exercise has been shown to produce significant improvements in key stroke rehabilitation outcomes, including functional movement, balance and cardiorespiratory fitness. Exercise programs have been shown to improve a variety of functional outcomes important for carrying out ADLs, including gait speed, gait endurance, Berg Balance Score, and 3-meter Timed Up and Go. Additionally, there is mounting evidence that aerobic exercise may improve cognitive recovery post-stroke. However, the research showing these effects has largely focused on exercise programs incorporated in a hospital or rehabilitation facility where patients are actively supervised by rehabilitation specialists. The American Heart Association recognizes that long-term and widely-applicable solutions for increasing exercise in post-stroke populations must hold the goal of exercise independence in the home and community settings.

Cycle ergometry, commonly known as an exercise bike, is a staple for stroke rehabilitation programs given its minimal fall risk and ability to produce moderate to vigorous intensity physical activity in participants. Exercise programs using cycle ergometry have been shown to produce all previously mentioned functional and cardiorespiratory improvements in stroke survivors, however, the translation of this effectiveness to the home-environment is unknown. Additionally, cycle ergometry may have smaller effects on functional mobility outcomes than walking interventions, forcing prescribing physicians and patients to choose between long-term improvement and reduced fall risk. One potential alternative or supplement to traditional aerobic exercise programs is exergaming, interventions which use physically active video games to engage participants in exercise. Exergames have been shown to be safe and produce moderate intensity physical activity levels in subacute and chronic stroke patients. Additionally, they have been shown to increase a variety of functional outcomes when added to standard post-stroke rehabilitation care, however, like aerobic exercise programs, previous research has focused on the supervised clinical setting, and it is unknown if they produce similar effects to aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Stroke greater than 3 months ago
* NIH stroke scale score less than 15

Exclusion Criteria:

* Other neurological impairments
* Medically unstable
* Inability to exercise
* Joint pain
* Heart failure or other heart arrythmias

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Average Gait Speed | baseline and 1 month
  Participants will walk as fast as possible on a 9-m runway 3 times, and the results will be averaged.

SECONDARY OUTCOMES:
VO2max | baseline and 1 month
  Maximal oxygen consumption (VO2max) will be determined by a breath by-breath measurement of VO2 with a Vmax Encore Metabolic System (CareFusion Corp, San Diego, CA), while participants perform a progressive ramped exercise test using an electronic-braked lower body cycle ergometer.
Timed up and GO | baseline and 1 month
  Participants will be asked to stand up from a seated position, walk 10 feet at a normal pace, then return to the chair and sit down. The examiner will time the procedure.
Berg Balance Scale | baseline and 1 month
  Participants will complete the 14 part Berg Balance test which requires them to complete basic functional movements that are each evaluated on a 4-point scale.
Cognition | baseline and 1 month
  Cognition will be assessed using a standardized, computerized test that is a part of the NIH Toolbox for Assessment of Neurological and Behavioral Function. It assesses various cognitive domains through simple, validated cognitive tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. Barbuto, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No